CLINICAL TRIAL: NCT02165176
Title: Pharmacokinetic and Pharmacodynamic Effects of Oral Cannabis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency); RTI International (Other)
Responsible Party: Principal Investigator, Ryan Vandrey, Associate Professor, Johns Hopkins University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00035394
Record Dates: First submitted 2014-06-12; First posted 2014-06-17 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Cannabis
Keywords: cannabis; toxicology; intoxication
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 10mg acute oral cannabis (Experimental): 10mg acute oral cannabis
  Interventions: Drug: Oral cannabis
- 25mg acute oral cannabis (Experimental): 25mg acute oral cannabis
  Interventions: Drug: Oral cannabis
- 50mg acute oral cannabis (Experimental): 50mg acute oral cannabis
  Interventions: Drug: Oral cannabis

INTERVENTIONS:
Drug: Oral cannabis

SUMMARY:
Few studies have been conducted to assess the pharmacokinetic and pharmacodynamic effects of orally consumed intact cannabis (e.g., cannabis-containing brownies). Careful analysis of oral cannabis dose effects on these parameters is required to determine the level and duration of biological cannabinoid exposure and associated subjective, cardiovascular and cognitive effects. In the present study we evaluated the detection of cannabinoids in oral fluid, plasma, hair, and urine for up to 9 days following consumption of oral cannabis (10mg, 25mg, or 50mg THC). The outcomes of the study will extend scientific knowledge about the behavioral pharmacology and toxicology of oral cannabis administration and can inform policies regarding clinical, workplace and roadside drug testing programs.

ELIGIBILITY:
Inclusion Criteria:

1. Have provided written informed consent
2. Be between the ages of 18 and 45
3. Be in good general health based on a physical examination, medical history, vital signs, 12-lead ECG and screening urine and blood tests
4. Test negative for recent cannabis use in urine at the screening visit (confirmed by GC/MS laboratory test) and at clinic admission
5. Test negative for other drugs of abuse, including alcohol at the screening visit and at clinic admission
6. Demonstrate ability to expectorate 3-5 mL of "native" oral fluid over a 5-minute period
7. Not be pregnant or nursing (if female). All females must have a negative serum pregnancy test at the screening visit and a negative urine pregnancy test at clinic admission.
8. Have a body mass index (BMI) in the range of 19 to 36 kg/m2
9. Have head hair that is at least 4 cm (approximately one and a half inches) in length on the back of the head.
10. Blood pressure at Screening Visit does not exceed a systolic blood pressure (SBP) of 150 mmHg or a diastolic blood pressure (DBP) of 90 mmHg
11. Have no allergies to any of the ingredients used to prepare cannabis brownies (chocolate, eggs, wheat, etc.).

Exclusion Criteria:

1. Non-medical use of psychoactive drugs other than, nicotine, alcohol, or caffeine 3 month prior to the Screening Visit;
2. History of or current evidence of significant medical or psychiatric illness judged by the investigator to put the participant at greater risk of experiencing an adverse event due to exposure or completion of other study procedures.
3. Use of an OTC, systemic or topical drug(s), herbal supplement(s), or vitamin(s) within 14 days of experimental sessions; which, in the opinion of the investigator or sponsor, will interfere with the study result or the safety of the subject.
4. Use of a prescription medication (with the exception of birth control prescriptions) within 14 days of experimental sessions; which, in the opinion of the investigator or sponsor, will interfere with the study result or the safety of the subject.
5. Use of hemp seeds or hemp oil in any form in the past 3 months.
6. Use of dronabinol (Marinol) within the past 6 months.
7. History of xerostomia (dry mouth), or the presence of mucositis, gum infection or bleeding, or other significant oral cavity disease or disorder that in the investigator's opinion may affect the collection of oral fluid samples.
8. History of clinically significant cardiac arrhythmias or vasospastic disease (e.g., Prinzmetal's angina).
9. Abnormal EKG result that in the investigator's opinion is clinically significant.
10. Enrolled in another clinical trial or have received any drug as part of a research study within 30 days prior to dosing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Blood THC | baseline and 0.2, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 22, 26, 30, 34, 46, 50, 54, 58, 70, 74, 78, 82, 94, 98, 102, 106, 118, 122, 126, and 130 hours post exposure
Urine THC-COOH | Baseline and 1, 2, 3, 4, 4-6 hours, 6-8 hours, 8-10 hours, 10-12 hours and then every 4 hours up until the 130 hour post exposure time point
Oral Fluid THC | baseline and 0.2, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 22, 26, 30, 34, 46, 50, 54, 58, 70, 74, 78, 82, 94, 98, 102, 106, 118, 122, 126, and 130 hours post exposure
Subjective rating of "Drug Effect" | baseline, immediately after exposure and 0.5, 1, 1.5, 2, 3, 4, 5, 6, and 8 hours post exposure
  Visual analog scale ratings of subjective intoxication

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Vandrey, PhD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins School of Medicine Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States